CLINICAL TRIAL: NCT06404268
Title: Facilitating Neuroplastic Changes of Acute Stroke Survivors With Severe Hemiplegia
Brief Title: Facilitating Neuroplastic Changes of Acute Stroke Survivors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Li-Qun Zhang, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00110205
Record Dates: First submitted 2024-05-01; First posted 2024-05-08 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: Stroke; Paraplegia; Acute
MeSH Terms: conditions — Stroke; Paraplegia | interventions — Muscle Stretching Exercises; Range of Motion, Articular

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with the study group and control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group - Wearable ankle robot rehab (Experimental): Wearable rehab robot with motor relearning with real-time feedback, passive stretching under intelligent control; Active movement training with robotic assistance
  Interventions: Device: Motor relearning training; Device: Passive stretching; Device: Gamed-based active movement training
- Control group - Limited wearable ankle robot rehab (Active Comparator): The same wearable robot used by the study group will be used for the control group but in a limited way: no motor relearning training under real-time feedback; passive movement in the joint middle range of motion instead of passive stretching; active movement training with no robotic assistance
  Interventions: Device: Passive movement; Device: Active movement training; Device: Ankle torque and motion measurement

INTERVENTIONS:
Device: Motor relearning training — Ankle motor control relearning training under real-time feedback
  Arms: Study group - Wearable ankle robot rehab
Device: Passive stretching — Passive stretching under intelligent robotic control
  Arms: Study group - Wearable ankle robot rehab
Device: Gamed-based active movement training — Active movement training through movement games with robotic assistance
  Arms: Study group - Wearable ankle robot rehab
Device: Passive movement — Passive movement in the joint middle range of motion
  Arms: Control group - Limited wearable ankle robot rehab
Device: Active movement training — Active movement training without robotic assistance
  Arms: Control group - Limited wearable ankle robot rehab
Device: Ankle torque and motion measurement — Ankle torque and motion measurement with no real-time feedback
  Arms: Control group - Limited wearable ankle robot rehab

SUMMARY:
This project will develop a wearable rehabilitation robot suitable for in-bed acute stage rehabilitation. It involves robot-guided motor relearning, passive and active motor-sensory rehabilitation early in the acute stage post-stroke including patients who are paralyzed with no motor output. The early acute stroke rehabilitation device will be evaluated in this clinical trial.

DETAILED DESCRIPTION:
Stroke survivors often experience loss of motor control and impaired function. Immediately after stroke, there is a time-limited window of heightened plasticity during which the greatest gains in recovery occur. Therefore, early intensive sensorimotor rehabilitation post-stroke is critical in improving functional outcomes and minimizing disability. However, acute stroke survivors often receive little active training to improve mobility during their hospital stay and they are left alone during most of the day. Especially for those acute patients with no voluntary motor output, active motor training might be even less, partly due to a lack of rehabilitation protocols to detect potential motor recovering signals sensitively and facilitate neuroplastic changes. To address this unmet clinical need, this project will develop a novel wearable rehabilitation robot suitable for in-bed acute stage rehabilitation with guided motor relearning, passive and active motor-sensory rehabilitation early in the acute stage post-stroke including patients who are paralyzed with no motor output. The early acute stroke rehabilitation device will be evaluated in this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Acute first time unilateral hemispheric stroke (hemorrhagic or ischemic stroke, 24 hours after admission to 1 month post-stroke at the start of the proposed treatment)
* Hemiplegia or hemiparesis
* 0≤Manual Muscle Testing (MMT)<=2
* Age 30-85
* Ankle impairments including stiff calf muscles and/or inadequate dorsiflexion

Exclusion Criteria:

* Medically not stable
* Associated acute medical illness that interferes with ability to training and exercise
* No impairment or very mild ankle impairment of ankle
* Severe cardiovascular problems that interfere with ability to perform moderate movement exercises
* Cognitive impairment or aphasia with inability to follow instructions
* Severe pain in legs
* Severe ankle contracture greater than 15° plantar flexion (when pushing ankle to dorsiflexion)
* Pressure ulcer, recent surgical incision or active skin disease with open wounds present below knee

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Lower Extremity (FMLE) | At the beginning and end of 3-week training, and 1 month after the treatment ends]
  The Fugl-Meyer Lower Extremity (FMLE) assessment is a measure of lower extremity (LE) motor and sensory impairments. The FMLE scale ranges from 0 to 34, with higher scores indicating better motor function.

SECONDARY OUTCOMES:
Active range of motion (AROM) | At the beginning and end of 3-week training, and 1 month after the treatment ends
  AROM will be measured in degrees in the ankle joint while subjects use the muscles to move the ankle.
Passive Range of Motion (PROM) will be measured in degrees in the ankle joint while the robot moves the ankle of the subject strongly. | At the beginning and end of 3-week training, and 1 month after the treatment ends
  Passive Range of Motion PROM will be measured in degrees in the ankle joint while the robot moves the ankle of the subject strongly.
Strength of the ankle flexor-extensor muscle will be measured in Newtons | At the beginning and end of 3-week training, and 1 month after the treatment ends
  Strength of the ankle flexor-extensor muscle will be measured in Newtons
Modified Ashworth Scale (MAS) | At the beginning and end of 3-week training, and 1 month after the treatment ends
  The Modified Ashworth Scale is the most widely used assessment tool to measure resistance to limb movement in a clinic setting. Scores range from 0-4, with 6 choices. 0 (0) - No increase in muscle tone; 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension; 1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM (range of movement); 2 (3) - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved; 3 (4) - Considerable increase in muscle tone passive, movement difficult; 4 (5) - Affected part(s) rigid in flexion or extension.
Berg Balance Scale | At the beginning and end of 3-week training, and 1 month after the treatment ends
  The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. The Berg balance scale ranges from 0 to 56. It is a 14-item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function.
10-meter Walk Test | At the beginning and end of 3-week training, and 1 month after the treatment ends
  The 10 Meter Walk Test is a performance measure used to assess walking speed in meters per second over a short distance at the beginning and end of 3-week training, and 1 month after the treatment ends. It can be employed to determine functional mobility and gait function.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Qun Zhang, Principal Investigator — University of Maryland
Locations (2):
- United States (2):
  - University of Maryland Baltimore, Baltimore, Maryland
  - UMROI, Baltimore, Maryland

REFERENCES:
- [Background] Zhang C, Huang MZ, Kehs GJ, Braun RG, Cole JW, Zhang LQ. Intensive In-Bed Sensorimotor Rehabilitation of Early Subacute Stroke Survivors With Severe Hemiplegia Using a Wearable Robot. IEEE Trans Neural Syst Rehabil Eng. 2021;29:2252-2259. doi: 10.1109/TNSRE.2021.3121204. Epub 2021 Nov 4. PMID 34665733
- [Background] Krakauer JW, Carmichael ST, Corbett D, Wittenberg GF. Getting neurorehabilitation right: what can be learned from animal models? Neurorehabil Neural Repair. 2012 Oct;26(8):923-31. doi: 10.1177/1545968312440745. Epub 2012 Mar 30. PMID 22466792
- [Background] Langhorne P, Bernhardt J, Kwakkel G. Stroke rehabilitation. Lancet. 2011 May 14;377(9778):1693-702. doi: 10.1016/S0140-6736(11)60325-5. PMID 21571152
- [Background] Nudo RJ, Milliken GW. Reorganization of movement representations in primary motor cortex following focal ischemic infarcts in adult squirrel monkeys. J Neurophysiol. 1996 May;75(5):2144-9. doi: 10.1152/jn.1996.75.5.2144. PMID 8734610
- [Background] Ren Y, Wu YN, Yang CY, Xu T, Harvey RL, Zhang LQ. Developing a Wearable Ankle Rehabilitation Robotic Device for in-Bed Acute Stroke Rehabilitation. IEEE Trans Neural Syst Rehabil Eng. 2017 Jun;25(6):589-596. doi: 10.1109/TNSRE.2016.2584003. Epub 2016 Jun 22. PMID 27337720
- [Background] Sanger TD, Delgado MR, Gaebler-Spira D, Hallett M, Mink JW; Task Force on Childhood Motor Disorders. Classification and definition of disorders causing hypertonia in childhood. Pediatrics. 2003 Jan;111(1):e89-97. doi: 10.1542/peds.111.1.e89. PMID 12509602
- [Background] Selles RW, Li X, Lin F, Chung SG, Roth EJ, Zhang LQ. Feedback-controlled and programmed stretching of the ankle plantarflexors and dorsiflexors in stroke: effects of a 4-week intervention program. Arch Phys Med Rehabil. 2005 Dec;86(12):2330-6. doi: 10.1016/j.apmr.2005.07.305. PMID 16344031
- [Background] Sukal-Moulton T, Clancy T, Zhang LQ, Gaebler-Spira D. Clinical application of a robotic ankle training program for cerebral palsy compared to the research laboratory application: does it translate to practice? Arch Phys Med Rehabil. 2014 Aug;95(8):1433-40. doi: 10.1016/j.apmr.2014.04.010. Epub 2014 May 2. PMID 24792141
- [Background] Waldman G, Yang CY, Ren Y, Liu L, Guo X, Harvey RL, Roth EJ, Zhang LQ. Effects of robot-guided passive stretching and active movement training of ankle and mobility impairments in stroke. NeuroRehabilitation. 2013;32(3):625-34. doi: 10.3233/NRE-130885. PMID 23648617
- [Background] Wu YN, Hwang M, Ren Y, Gaebler-Spira D, Zhang LQ. Combined passive stretching and active movement rehabilitation of lower-limb impairments in children with cerebral palsy using a portable robot. Neurorehabil Neural Repair. 2011 May;25(4):378-85. doi: 10.1177/1545968310388666. Epub 2011 Feb 22. PMID 21343525
- [Background] Wu YN, Ren Y, Goldsmith A, Gaebler D, Liu SQ, Zhang LQ. Characterization of spasticity in cerebral palsy: dependence of catch angle on velocity. Dev Med Child Neurol. 2010 Jun;52(6):563-9. doi: 10.1111/j.1469-8749.2009.03602.x. Epub 2010 Jan 28. PMID 20132137
- [Background] Xerri C, Merzenich MM, Peterson BE, Jenkins W. Plasticity of primary somatosensory cortex paralleling sensorimotor skill recovery from stroke in adult monkeys. J Neurophysiol. 1998 Apr;79(4):2119-48. doi: 10.1152/jn.1998.79.4.2119. PMID 9535973
- [Background] Yang CY, Guo X, Ren Y, Kang SH, Zhang LQ. Position-dependent, hyperexcitable patellar reflex dynamics in chronic stroke. Arch Phys Med Rehabil. 2013 Feb;94(2):391-400. doi: 10.1016/j.apmr.2012.09.029. Epub 2012 Oct 11. PMID 23063880
- [Background] Zhang LQ, Chung SG, Ren Y, Liu L, Roth EJ, Rymer WZ. Simultaneous characterizations of reflex and nonreflex dynamic and static changes in spastic hemiparesis. J Neurophysiol. 2013 Jul;110(2):418-30. doi: 10.1152/jn.00573.2012. Epub 2013 May 1. PMID 23636726
- [Background] Zhang LQ, Rymer WZ. Reflex and intrinsic changes induced by fatigue of human elbow extensor muscles. J Neurophysiol. 2001 Sep;86(3):1086-94. doi: 10.1152/jn.2001.86.3.1086. PMID 11535659
- [Background] Zhang LQ, Wang G, Nishida T, Xu D, Sliwa JA, Rymer WZ. Hyperactive tendon reflexes in spastic multiple sclerosis: measures and mechanisms of action. Arch Phys Med Rehabil. 2000 Jul;81(7):901-9. doi: 10.1053/apmr.2000.5582. PMID 10896002
- [Background] Zhao H, Wu YN, Hwang M, Ren Y, Gao F, Gaebler-Spira D, Zhang LQ. Changes of calf muscle-tendon biomechanical properties induced by passive-stretching and active-movement training in children with cerebral palsy. J Appl Physiol (1985). 2011 Aug;111(2):435-42. doi: 10.1152/japplphysiol.01361.2010. Epub 2011 May 19. PMID 21596920
- [Background] Albert SJ, Kesselring J. Neurorehabilitation of stroke. J Neurol. 2012 May;259(5):817-32. doi: 10.1007/s00415-011-6247-y. Epub 2011 Oct 1. PMID 21964750
- [Background] Bernhardt J, Chan J, Nicola I, Collier JM. Little therapy, little physical activity: rehabilitation within the first 14 days of organized stroke unit care. J Rehabil Med. 2007 Jan;39(1):43-8. doi: 10.2340/16501977-0013. PMID 17225037
- [Background] Bernhardt J, Dewey H, Thrift A, Donnan G. Inactive and alone: physical activity within the first 14 days of acute stroke unit care. Stroke. 2004 Apr;35(4):1005-9. doi: 10.1161/01.STR.0000120727.40792.40. Epub 2004 Feb 26. PMID 14988574
- [Background] Chung SG, van Rey E, Bai Z, Rymer WZ, Roth EJ, Zhang LQ. Separate quantification of reflex and nonreflex components of spastic hypertonia in chronic hemiparesis. Arch Phys Med Rehabil. 2008 Apr;89(4):700-10. doi: 10.1016/j.apmr.2007.09.051. PMID 18374001
- [Background] Chung SG, Van Rey E, Bai Z, Roth EJ, Zhang LQ. Biomechanic changes in passive properties of hemiplegic ankles with spastic hypertonia. Arch Phys Med Rehabil. 2004 Oct;85(10):1638-46. doi: 10.1016/j.apmr.2003.11.041. PMID 15468024
- [Background] Chen K, Wu YN, Ren Y, Liu L, Gaebler-Spira D, Tankard K, Lee J, Song W, Wang M, Zhang LQ. Home-Based Versus Laboratory-Based Robotic Ankle Training for Children With Cerebral Palsy: A Pilot Randomized Comparative Trial. Arch Phys Med Rehabil. 2016 Aug;97(8):1237-43. doi: 10.1016/j.apmr.2016.01.029. Epub 2016 Feb 20. PMID 26903143
- [Background] Quality Standards Subcommittee of the American Academy of Neurology and the Practice Committee of the Child Neurology Society; Delgado MR, Hirtz D, Aisen M, Ashwal S, Fehlings DL, McLaughlin J, Morrison LA, Shrader MW, Tilton A, Vargus-Adams J. Practice parameter: pharmacologic treatment of spasticity in children and adolescents with cerebral palsy (an evidence-based review): report of the Quality Standards Subcommittee of the American Academy of Neurology and the Practice Committee of the Child Neurology Society. Neurology. 2010 Jan 26;74(4):336-43. doi: 10.1212/WNL.0b013e3181cbcd2f. PMID 20101040
- [Background] Gao F, Grant TH, Roth EJ, Zhang LQ. Changes in passive mechanical properties of the gastrocnemius muscle at the muscle fascicle and joint levels in stroke survivors. Arch Phys Med Rehabil. 2009 May;90(5):819-26. doi: 10.1016/j.apmr.2008.11.004. PMID 19406302
- [Background] Gao F, Ren Y, Roth EJ, Harvey R, Zhang LQ. Effects of repeated ankle stretching on calf muscle-tendon and ankle biomechanical properties in stroke survivors. Clin Biomech (Bristol). 2011 Jun;26(5):516-22. doi: 10.1016/j.clinbiomech.2010.12.003. Epub 2011 Jan 6. PMID 21211873
- [Background] Gao F, Zhang LQ. Altered contractile properties of the gastrocnemius muscle poststroke. J Appl Physiol (1985). 2008 Dec;105(6):1802-8. doi: 10.1152/japplphysiol.90930.2008. Epub 2008 Oct 23. PMID 18948443
- [Background] Jenkins WM, Merzenich MM. Reorganization of neocortical representations after brain injury: a neurophysiological model of the bases of recovery from stroke. Prog Brain Res. 1987;71:249-66. doi: 10.1016/s0079-6123(08)61829-4. No abstract available. PMID 3588947